CLINICAL TRIAL: NCT04814537
Title: A Trial to Determine the Optimal Bupivacaine Dose for Initiation of Labor Epidural Pain Relief
Brief Title: Optimal Bupivacaine Dose for Initiation of Labor Epidural Techniques
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Lawrence Ching Tsen, Associate Professor of Anesthesia, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020P003241
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Labor Pain; Analgesia
Keywords: Dural Puncture Epidural Technique; Epidural Technique; Neuraxial Labor Analgesia; Bupivacaine; Local Anesthetic Agent
MeSH Terms: conditions — Labor Pain; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial Using Biased Coin Design to Determine Effective Dose for 90% (ED90) of Subjects
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The biased-coin allocation after each successful response will be implemented by flipping a virtual biased coin (10% vs. 90% probability of randomizing the next patient to the lower vs. same dose than received by the last patient with the same epidural technique) using R statistical software (R Foundation for Statistical Computing, Vienna, Austria). Care Provider (Clinical Anesthesiologist) will administer the identified dose, then summon blinded observer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dural Puncture Epidural Technique (Experimental): Laboring women receiving the Dural Puncture Epidural (DPE) Technique with dose of Bupivacaine 0.25% diluted to 20 mL with isotonic sterile 0.9% saline. The first subject in the DPE group will receive an initial dose of bupivacaine 25 mg, with an endpoint being the achievement of an NRS < 3 at 30 min. Subsequent patients are administered bupivacaine doses determined by the response of the previous subject, as per the biased coin method. The subsequent up and down interval doses are bupivacaine 2.5 mg (1 mL) increments, with an anticipated dose range from 20 mg to 40 mg.
  Interventions: Drug: Bupivacaine Hydrochloride
- Epidural Technique (Active Comparator): Laboring women receiving the Conventional Epidural Technique (EPL) with dose of Bupivacaine 0.25% diluted to 20 mL with isotonic sterile 0.9% saline. The first subject in the EPL group will receive an initial dose of bupivacaine 25 mg, with an endpoint being the achievement of an NRS < 3 at 30 min. Subsequent patients are administered bupivacaine doses determined by the response of the previous subject, as per the biased coin method. The subsequent up and down interval doses are bupivacaine 2.5 mg (1 mL) increments, with an anticipated dose range from 20 mg to 40 mg.
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — Local Anesthetic Agent
  Other Names: Marcaine

SUMMARY:
To estimate the dose of bupivacaine required to achieve initial effective comfort in 90% of patients (ED90) via the epidural (DPE or EPL) technique in women undergoing labor.

DETAILED DESCRIPTION:
The primary objective of our study is to use a biased coin up-down allocation methodology to estimate the dose of bupivacaine required to achieve initial effective comfort in 90% of patients (ED90) via the epidural (DPE or EPL) technique in women undergoing labor induction or augmentation; we hypothesize that we will be able to determine the ED90 of bupivacaine for each technique with adequate precision to inform the optimal doses.

ELIGIBILITY:
Inclusion Criteria:

1. Parturient with no major co-morbidities
2. Singleton, vertex gestation at term (37-42 weeks)
3. Less than or equal to 5 cm dilation
4. Desire to receive epidural labor analgesia
5. Numerical Rating Scale greater or equal to 5 (NRS 0-10, where 0 = no pain, and 10 = worst pain imaginable), at time of epidural labor analgesia request.

Exclusion Criteria:

1. Current or historical evidence of clinically significant disease or condition, including diseases of pregnancy (i.e preeclampsia, gestational diabetes)
2. Any contraindication to the administration of an epidural technique
3. History of hypersensitivity or idiosyncratic reaction to an amide local anesthetic agent
4. Current or historical evidence of a disease which may result in the risk of a cesarean delivery (i.e. history of uterine rupture). NB: Exception-trial of labor after cesarean delivery (TOLAC) will be eligible.
5. Evidence of anticipated fetal anomalies

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant Women
Enrollment: 100 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
Verbal Numerical Rating Score (0-10, with higher scores meaning more pain); goal with analgesia is < 3/10 | 30 minutes
  Pain Score (0=no pain, 10= worst pain imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Tsen, MD, Principal Investigator — Associate Professor in Anesthesiology, Harvard Medical School
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ngan Kee WD, Ng FF, Khaw KS, Lee A, Gin T. Determination and comparison of graded dose-response curves for epidural bupivacaine and ropivacaine for analgesia in laboring nulliparous women. Anesthesiology. 2010 Aug;113(2):445-53. doi: 10.1097/ALN.0b013e3181bdf9da. PMID 20613484
- [Result] Benhamou D, Ghosh C, Mercier FJ. A randomized sequential allocation study to determine the minimum effective analgesic concentration of levobupivacaine and ropivacaine in patients receiving epidural analgesia for labor. Anesthesiology. 2003 Dec;99(6):1383-6. doi: 10.1097/00000542-200312000-00022. PMID 14639153
- [Result] Chau A, Bibbo C, Huang CC, Elterman KG, Cappiello EC, Robinson JN, Tsen LC. Dural Puncture Epidural Technique Improves Labor Analgesia Quality With Fewer Side Effects Compared With Epidural and Combined Spinal Epidural Techniques: A Randomized Clinical Trial. Anesth Analg. 2017 Feb;124(2):560-569. doi: 10.1213/ANE.0000000000001798. PMID 28067707
- [Derived] Maeda A, Villela-Franyutti D, Lumbreras-Marquez MI, Murthy A, Fields KG, Justice S, Tsen LC. Labor Analgesia Initiation With Dural Puncture Epidural Versus Conventional Epidural Techniques: A Randomized Biased-Coin Sequential Allocation Trial to Determine the Effective Dose for 90% of Patients of Bupivacaine. Anesth Analg. 2024 Jun 1;138(6):1205-1214. doi: 10.1213/ANE.0000000000006691. Epub 2023 Oct 12. PMID 37824436